CLINICAL TRIAL: NCT00113451
Title: Radial Artery Bypass Graft Study of Tromsø
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Other Study IDs: SFP-091-03; P-REK Nord 82/2003
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Coronary Arteriosclerosis; Myocardial Infarction
Keywords: radial artery; angina pectoris; infarction; bypass; angiography
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina Pectoris; Infarction

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to answer, among others, the following questions: 1) What are the outcomes when using the radial artery as a bypass graft in coronary artery bypass surgery (CABG)? 2) Can multidetector computed tomography (CT) be used to reliably evaluate coronary artery bypass graft patency?

DETAILED DESCRIPTION:
Radial arteries have been used as aortocoronary conduits with varying results. The study is based on the first 119 patients operated with this graft at our institution, aiming to answer the following questions:

1. What is the short-term patency (2-3 years) of radial artery bypass grafts in CABG (comparisons are made with saphenous veins and internal thoracic artery grafts)?
2. What complications occur and what in what frequency?
3. What are the clinical outcomes and patient satisfaction after using radial arteries in CABG? (n=119 pt.)
4. Can multidetector CT be used to reliably evaluate coronary artery bypass graft patency? (n=45 pt.)

Methods: Questionnaires, record review, coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Operated with radial artery coronary bypass at our department during April 2001 - October 2004
* Written informed consent

Exclusion Criteria:

* For the angiography procedures, standard contraindications are adhered to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119
Dates: Start 2004-01; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- The University Hospital of North Norway, Tromsø, Tromsø, Norway